CLINICAL TRIAL: NCT00861926
Title: 48-week,Multinational,Randomized,Double-blind,2-parallel Groups,Comparing the Efficacy of Foster for Maintenance and Reliever Versus Fixed-dose Foster for Maintenance Plus Salbutamol as Reliever in Asthmatics >=18 Years of Age
Brief Title: Study Comparing Foster Efficacy Maintenance and Reliever Versus Foster Maintenance + Salbutamol Reliever in Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-0804-PR-0034
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Maintenance and Reliever Treatments
MeSH Terms: conditions — Asthma | interventions — Albuterol; Beclomethasone; Formoterol Fumarate; Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beclometasone/formoterol (100/6 µg) (Experimental): Foster : fixed combination of BDP extrafine 100 µg plus formoterol fumarate 6 µg administered via a pMDI standard actuator
  Interventions: Drug: beclometasone /formoterol
- salbutamol (Active Comparator): Ventolin : salbutamol sulphate 100 µg per metered dose
  Interventions: Drug: Ventolin

INTERVENTIONS:
Drug: Ventolin — Ventolin : salbutamol sulfate 100µg
  Arms: salbutamol
Drug: beclometasone /formoterol — BDP 100µg/FF 6µg, 1 inhalation bid
  Other Names: Foster
  Arms: Beclometasone/formoterol (100/6 µg)

SUMMARY:
Double-blind, multinational, multicentre, randomized, 2-arm parallel-group study

DETAILED DESCRIPTION:
To compare efficacy of Foster as maintenance therapy plus additional inhalations as reliever with Foster as maintenance plus salbutamol as reliever in asthmatics

ELIGIBILITY:
Inclusion Criteria:

* Written signed and dated informed consent obtained.
* Male or female patients aged ≥ 18 years.
* A positive reversibility test
* Patients who experienced at least one severe exacerbation in the 12 months before entry (but not in the last month)
* Using inhaled corticosteroids (ICS) in monotherapy or using ICS in a fixed or free combination with long acting beta2 agonists (LABA) at a constant dose for two months before screening visit
* Not fully controlled asthmatics (which means partly controlled or/and uncontrolled patients according to GINA guidelines 2007) in the last month before screening visit
* Forced expiratory volume in the first second (FEV1) ≥ 60% of predicted for the patient normal value.
* Non smokers or ex-smokers

Exclusion Criteria:

* Pregnant or nursing (lactating) women. Women of child-bearing potential UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or are using one or more of acceptable methods of contraception
* Body Mass Index (BMI) > 34 kg/m2.
* Patient with lower respiratory tract infections affecting the patient's asthma within 30 days of the screening visit.
* Use of systemic steroids in the last month.
* Patients with other lung diseases such as COPD, cystic fibrosis, interstitial lung diseases or any other clinically or functionally significant lung disorder.
* Patients who have an uncontrolled respiratory, haematological, immunologic, renal, neurologic, hepatic, endocrinal or other disease.
* Clinically relevant laboratory abnormalities
* Patients who have an abnormal QTcF interval value
* Intolerance or contra-indication to treatment with beta2-agonists and/or ICS or allergy to any component of the study treatments.
* Patients treated with slow-release corticosteroids in the 3 months prior to screening visit.
* Patients being treated with anti-IgE antibodies.
* Patients treated with LABA or ICS/LABA fixed combination in the 24h before screening visit
* Severe asthma exacerbation in the last month before screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2079 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation | At each clinic visit

SECONDARY OUTCOMES:
Number of severe asthma exacerbations Number of hospitalization Asthma symptoms Rescue medication LFTs | At each clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, Professor, Principal Investigator — Universita degli Studi di Ferrara
Locations (1):
- Pr Papi, Ferrara, Italy

REFERENCES:
- [Result] Papi A, Corradi M, Pigeon-Francisco C, Baronio R, Siergiejko Z, Petruzzelli S, Fabbri LM, Rabe KF. Beclometasone-formoterol as maintenance and reliever treatment in patients with asthma: a double-blind, randomised controlled trial. Lancet Respir Med. 2013 Mar;1(1):23-31. doi: 10.1016/S2213-2600(13)70012-2. Epub 2013 Mar 4. PMID 24321801
- [Derived] Morjaria JB, Rigby AS, Morice AH. Symptoms and exacerbations in asthma: an apparent paradox? Ther Adv Chronic Dis. 2019 Oct 24;10:2040622319884387. doi: 10.1177/2040622319884387. eCollection 2019. PMID 31695864
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2008-004671-22